CLINICAL TRIAL: NCT03113006
Title: The Individually-Marked Panretinal Laser phoTocoagulation for Proliferative Diabetic Retinopathy Study: IMPETUS 2018 - TREAT
Brief Title: The Individually-Marked Panretinal Laser phoTocoagulation for Proliferative Diabetic Retinopathy Study (TREAT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other); Velux Fonden (Other)
Responsible Party: Principal Investigator, Anna Stage Vergmann, Ph. D. student, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-20160168
Record Dates: First submitted 2017-03-24; First posted 2017-04-13 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Proliferative Diabetic Retinopathy; PDR; Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Panretinal Photocoagulation (Active Comparator): Localized to all four retinal quadrants.
  Interventions: Procedure: Panretinal Photocoagulation
- Individ. Panretinal Photocoagulation (Experimental): Localized to only the affected quadrants.
  Interventions: Procedure: Panretinal Photocoagulation

INTERVENTIONS:
Procedure: Panretinal Photocoagulation — Panretinal laser treatment of the retina in patients with proliferative diabetic retinopathy.
  Other Names: PRP

SUMMARY:
Background Diabetic eye disease is the most frequent complication among the 320,000 Danes with diabetes. The formation of new vessels (PDR) in the inner part of the eye (retina) is a feared complication and a leading cause of blindness, since these vessels are fragile and often cause bleeding within the eye. Peripheral retinal laser treatment (PRP) halves the risk of blindness, but often comes with a high prize. The peripheral part of the retina is responsible for the visual field and the night vision, and PRP limits these abilities (i.e. loss of driving license).

The technique of PRP has principally been the same for the past 40 years with standard treatment given for all patients. With this one size fits all approach, a substantial number of patients will either be treated too much or too little. Too little treatment is inefficient, and disease progression may occur. Excessive treatment may cause side effects like loss of visual fields and decreased night vision. Therefore, it is important to test if treatment can be applied on an individual basis to give high efficacy treatment with minimal side effects.

IMPETUS 2018 - TREAT is the second of two studies aimed at making an individual design for retinal laser treatment. In IMPETUS 2018 - DETECT the investigators demonstrated that non-invasive examinations of the oxygen level and measurements of the retinal vascular tree provide important information of individual treatment response. For instance, if standard PRP led to three per cent higher retinal oxygen saturation, there was a 4-fold risk of disease progression despite treatment. Hence, such a patient would benefit from more treatment to avoid blindness. With these observations at hand, the investigators want to compare a less invasive treatment (individualized laser treatment) against the standard PRP.

Another essential aspect in the treatment of PDR is to be able to give the right diagnosis and to evaluate the efficacy of laser treatment. So far, this has been performed by fluorescein angiography. However, this examination are highly person-dependent and unpleasant to patients, and a more objective approach is needed. Optical coherent tomography angiography (OCT-A) is a quick, noninvasive scanning of the retina which is ideal to visualize moving objects like blood within the retinal vessels. The method has been successfully implemented in a number of retinal diseases, but it has never been validated in PDR.

Standard PRP is often performed in 3-4 sessions. However, it may be painful, and patients sometimes choose not to complete all sessions after the initial treatment has been given. There is insufficient knowledge of the patient-barriers to treatment, and it is important to address these in an individualized treatment design.

Aim In this 6-month 1:1 randomized, prospective study the investigators want to investigate 1) whether individualized retinal laser treatment compared with standard PRP has the same efficacy but less side effects, 2) whether OCT-A can be used as an objective marker for disease activity, and 3) to obtain a better understanding of patient-reported barriers to standard laser treatment PRP and whether these can be addressed with personalized retinal laser treatment.

Setup Fifty eight consecutively recruited patients (1 May 2017 - 30 April 2018) with newly diagnosed PDR referred to the Department of Ophthalmology, OUH, and randomly assigned to standard PRP (n=29) or individualized laser treatment (n=29).

Intervention Standard laser treatment is performed in all four quadrants of the retina. Individualized laser treatment is only performed in the part(s) of the retina with proliferation(s).

Both treatments are carried out at baseline (BL), and additional treatment is given at month three (M3) and/or (M6), if necessary.

Investigations Retinal digital images, fluorescein angiography, OCT-A (BL, M3, M6). Test of visual fields, dark adaptation and quality of life (BL, M6). Semi-structured interview will be performed with five patients who have received PRP in one eye and individualized laser treatment in the other eye. This will address treatment experience, potential barriers to treatment, etc.

What to measure:

Differences in need for retreatment, night blindness, visual fields, visual acuity, bleeding in the eye, surgery, and quality of life between the groups.

DETAILED DESCRIPTION:
Introduction Diabetes mellitus is an epidemic disorder, which in Denmark alone is affecting 320,000 patients. Diabetic retinopathy (DR) is the most frequent long term complication to diabetes mellitus (1) and a feared cause of severe vision loss and blindness (2).

Proliferative diabetic retinopathy (PDR) is the major cause of severe visual loss. Lack of oxygen to the retina (retinal ischemia) results in up-regulation of, in particular, the growth factor vascular endothelial growth factor (VEGF) (3) followed by compensatory retinal proliferations. The neovasculature is fragile and often leads to vitreous hemorrhages or retinal detachment which makes the patient at high risk of irreversible vision loss (4).

In 1976 it was shown that patients with severe PDR can halve the risk of severe vision loss by peripheral retinal laser treatment (photocoagulation panretinal, PRP) (5). This treatment reduces the retina's oxygen demand, which makes the VEGF concentration decrease and the proliferations shrink (5).

PRP has largely been the same for the last 40 years. The standard treatment is basically the same for all patients (4 + 6), which leads to some patients being either over or under treated. If treatment is inadequate, patients are in risk of disease progression and thus difficult vision loss (7). On the other hand, the treatment may cause side effects in the form of loss of visual field (8-9), night vision loss (10) and accumulation of fluid in the eye's macula (diabetic macular edema) (11).

This study is a continuum of the clinical project IMPETUS 2018 - DETECT, which aimed to identify the factors that were important for a successful PRP treatment of PDR. In the study the investigators prospectively followed 65 patients with newly diagnosed PDR. All patients received baseline navigated PRP, as in Scandinavia only offered at Odense University Hospital (OUH). Navigated panretinal laser with a Navilas® laser ensures optimized treatment (12), shorter treatment (13) and increased patient comfort (12-14). Treatment effect was investigated at month three and six, and if necessary, treatment was supplied. All the patients venous retinal oxygen saturation was measured to study whether this had any therapeutic value.

The investigators observed that the retinal oxygen saturation was a strong predictor of treatment response. Compared to patients whose disease was slowed down after treatment, patients with progression three months after PRP had an increase in the venous retinal oxygen saturation (+ 4.1% vs. -1.8%, p = 0.02). Patients with an increase of at least 3.0% in venous retinal oxygen saturation had 4.0 times greater risk of disease progression than patients who were below this threshold (15). This observation is in line with another Danish study, which demonstrated that worsening of DR causes increased venous retinal oxygen saturation (16). By measuring if this increase in venous retinal oxygen saturation has slowed down, one can assess whether PRP treatment is sufficient.

PDR is traditionally perceived as an ischemic disease, which initially affects the entire retina. In our above mentioned study the investigators were able to confirm the results regarding the venous retinal oxygen saturation in the affected segment of the retina, in 24 of the patients in the study, who had only one peripheral proliferation. In these patients the oxygen saturation was increased with disease progression (+ 3.9% vs. -1.5%, p = 0.04). This indicates that the focal hypoxia are more important than previously thought, and thus the local treatment of the diseased area may be a treatment option that reduces the processing volume, thereby minimizing potential side effects.

Retinal proliferations are fragile and often leak contrast fluid. When initiating the study, the investigators expected the leakage of fluorescein over time would be the optimal method to assess disease activity, but had to realize that this method was difficult to objectify (17). As an alternative to this objective evaluation, it is possible to observe the structural conditions at the interface between the retina and vitreous body (18), but technological limitations have so far prevented the possibility of repeated evaluations of the same lesion over time. Optical coherency tomography (OCT)-angiography is, however, a new method that can visualize retinal structures and potential development of these in detail (19).

Purpose In a six-month randomized, prospective study of patients with newly diagnosed PDR the investigators want to investigate 1) whether individualized PRP compared with standard PRP has the same efficacy but less side effects and 2) whether OCT angiography can be used as a marker for disease activity in PDR.

Hypothesis The investigators expect that 1) individualized PDR provides the same effect but fewer side effects and better quality of life than traditional PDR, and 2) OCT angiography has better sensitivity and specificity than wide field fluorescein angiography (FA) for the evaluation of disease activity by PDR.

Methods

Setup:

* Six-months 1: 1 randomized, prospective study.
* 58 consecutively recruited patients with newly diagnosed PDR at the Department of Ophthalmology, University Hospital, included in the period 1 March 2017 to 28 February 2018.
* Patients will be randomized to either 1) standard PRP with Navilas® (n = 29) or individualized PRP with Navilas® (n = 29). To ensure the same degree of ischemic disease, the two groups are balanced in relation to the number of retinal quadrants with proliferations.

Intervention:

* Standard PRP: localized to all four retinal quadrants.
* Individualized PRP: localized to the affected quadrants.
* Both treatments are carried out at baseline (BL) and supplemented if there is increasing disease activity at month three (M3) and / or month six (M6).
* Indications for additional treatment:
* Progression of PDR in the form of subjective growing lesion (assessed by ophthalmoscopy and wide field fundus photo) or increasing leakage wide field FA (M3 or M6).
* Progression of PDR in terms of objectively progressive lesion (≥10% from BL) measured by spectral domain (SD) OCT or OCT angiography (M3 or M6).
* Increase in venous retinal oxygen saturation of at least + 3,0% between BL and M3.

Investigations:

* Demographics: age, sex, type of diabetes, diabetes duration, smoking, drugs (BL).
* Objectively: Blood pressure, height, weight (BL).
* Blood samples: HbA1c, total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides, P creatinine, eGFR (BL, M3, M6).
* Visual acuity (Best Corrected Early Treatment Diabetic Retinopathy Study standard) (BL, M3, M6).
* Intraocular pressure (BL, M3, M6).
* SD-OCT (Topcon 3D OCT 2000): macula and area(s) with PDR (BL, M3, M6).
* OCT angiography (Topcon DRI OCT Triton): region(s) with PDR (BL, M3, M6).
* Wide field fundus photo and FA (Optos) (BL, M3, M6).
* Retinal oximetry (Oxymap T1) (BL, M3, M6).
* Dark-adaptation (Goldmann-weeker adaptometer) (BL, M6).
* Perimetry (Humphrey 30-2) (BL, M6).
* Selected components of quality of life questionnaire (Danish translation of Visual Function Questionnaire-25) (BL, M6).

Endpoints

Primary:

* Need for retreatment between the groups (M3 and M6).
* Loss of visual fields between the groups (from BL to M6).
* Change in dark adaptation between the groups (from BL to M6).
* Sensitivity and specificity of OCT angiography as an expression of disease activity in PDR (BL, M3 and M6).

Secondary:

* Change in visual acuity between the groups (from BL to M6).
* Difference in proportion with the development of vitreous haemorrhage between the groups (from BL to M6).
* Need for surgical removal of the vitreous between the groups (from BL to M6)
* Change in quality of life between the groups (from BL to M6).

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus.
* Newly diagnosed, untreated PDR in one eye (the possibility of inclusion of both eyes by bilateral PDR).

Exclusion Criteria:

* Diabetic macular edema in the affected eye.
* Age <18 years.
* Pregnancy.
* Ambiguities in refracting media on topical eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-08-27 (Actual)

PRIMARY OUTCOMES:
Need for retreatment between the groups | At month 3 and 6
  Change in the progression of PDR, hence the difference in the need for retreatment between the standard laser treatment group vs. the individualized laser treatment group.
Loss of visual fields between the groups | From baseline to month 6
  Loss of visual field between the standard laser treatment group vs. the individualized laser treatment group.
Change in dark adaptation between the groups | From baseline to month 6
  Change in dark adaptation between the standard laser treatment group vs. the individualized laser treatment group.
Sensitivity and specificity of OCT angiography as an expression of disease activity in PDR | At month 6
  The specificity and sensitivity of OCT-A in detecting progression in PDR

SECONDARY OUTCOMES:
Change in visual acuity between the groups | From baseline to month 6
  Change in visual acuity between the standard laser treatment group vs. the individualized laser treatment group.
Difference in proportion with the development of vitreous haemorrhage between the groups | From baseline to month 6
  Difference in proportion with the development of vitreous haemorrhage between the standard laser treatment group vs. the individualized laser treatment group.
Need for surgical removal of the vitreous between the groups | From baseline to month 6
  Need for surgical removal of the vitreous between the standard laser treatment group vs. the individualized laser treatment group.
Change in quality of life between the groups | From baseline to month 6
  Change in quality of life between the standard laser treatment group vs. the individualized laser treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Anna S Vergmann, M.D., Principal Investigator — Odense University Hospital
Locations (1):
- The Department of Ophthalmology, Odense University Hospital, Odense, The Region of Southern Denmarj, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grauslund J, Green A, Sjolie AK. Prevalence and 25 year incidence of proliferative retinopathy among Danish type 1 diabetic patients. Diabetologia. 2009 Sep;52(9):1829-35. doi: 10.1007/s00125-009-1450-4. Epub 2009 Jul 12. PMID 19593541
- [Background] Grauslund J, Green A, Sjolie AK. Blindness in a 25-year follow-up of a population-based cohort of Danish type 1 diabetic patients. Ophthalmology. 2009 Nov;116(11):2170-4. doi: 10.1016/j.ophtha.2009.04.043. Epub 2009 Sep 10. PMID 19744716
- [Background] Stefansson E. Ocular oxygenation and the treatment of diabetic retinopathy. Surv Ophthalmol. 2006 Jul-Aug;51(4):364-80. doi: 10.1016/j.survophthal.2006.04.005. PMID 16818083
- [Background] Photocoagulation treatment of proliferative diabetic retinopathy. Clinical application of Diabetic Retinopathy Study (DRS) findings, DRS Report Number 8. The Diabetic Retinopathy Study Research Group. Ophthalmology. 1981 Jul;88(7):583-600. PMID 7196564
- [Background] Preliminary report on effects of photocoagulation therapy. The Diabetic Retinopathy Study Research Group. Am J Ophthalmol. 1976 Apr;81(4):383-96. doi: 10.1016/0002-9394(76)90292-0. PMID 944535
- [Background] Early photocoagulation for diabetic retinopathy. ETDRS report number 9. Early Treatment Diabetic Retinopathy Study Research Group. Ophthalmology. 1991 May;98(5 Suppl):766-85. PMID 2062512
- [Background] Bandello F, Brancato R, Menchini U, Virgili G, Lanzetta P, Ferrari E, Incorvaia C. Light panretinal photocoagulation (LPRP) versus classic panretinal photocoagulation (CPRP) in proliferative diabetic retinopathy. Semin Ophthalmol. 2001 Mar;16(1):12-8. doi: 10.1076/soph.16.1.12.4223. PMID 15487693
- [Background] Fong DS, Girach A, Boney A. Visual side effects of successful scatter laser photocoagulation surgery for proliferative diabetic retinopathy: a literature review. Retina. 2007 Sep;27(7):816-24. doi: 10.1097/IAE.0b013e318042d32c. PMID 17891003
- [Background] Pahor D. Visual field loss after argon laser panretinal photocoagulation in diabetic retinopathy: full- versus mild-scatter coagulation. Int Ophthalmol. 1998;22(5):313-9. doi: 10.1023/a:1006367029134. PMID 10826550
- [Background] Pender PM, Benson WE, Compton H, Cox GB. The effects of panretinal photocoagulation on dark adaptation in diabetics with proliferative retinopathy. Ophthalmology. 1981 Jul;88(7):635-8. doi: 10.1016/s0161-6420(81)34977-x. PMID 7196565
- [Background] Ferris FL 3rd, Podgor MJ, Davis MD. Macular edema in Diabetic Retinopathy Study patients. Diabetic Retinopathy Study Report Number 12. Ophthalmology. 1987 Jul;94(7):754-60. doi: 10.1016/s0161-6420(87)33526-2. PMID 3658347
- [Background] Chhablani J, Mathai A, Rani P, Gupta V, Arevalo JF, Kozak I. Comparison of conventional pattern and novel navigated panretinal photocoagulation in proliferative diabetic retinopathy. Invest Ophthalmol Vis Sci. 2014 May 1;55(6):3432-8. doi: 10.1167/iovs.14-13936. PMID 24787564
- [Background] Chhablani J, Sambhana S, Mathai A, Gupta V, Arevalo JF, Kozak I. Clinical efficacy of navigated panretinal photocoagulation in proliferative diabetic retinopathy. Am J Ophthalmol. 2015 May;159(5):884-9. doi: 10.1016/j.ajo.2015.02.006. Epub 2015 Feb 19. PMID 25703478
- [Background] Inan UU, Polat O, Inan S, Yigit S, Baysal Z. Comparison of pain scores between patients undergoing panretinal photocoagulation using navigated or pattern scan laser systems. Arq Bras Oftalmol. 2016 Feb;79(1):15-8. doi: 10.5935/0004-2749.20160006. PMID 26840160
- [Background] Torp TL, Kawasaki R, Wong TY, Peto T, Grauslund J. Improvement in retinal venous oxygen saturation after panretinal photocoagulation is predictive of progression of proliferative diabetic retinopathy. ARVO, 2016;6356-C0143.
- [Background] Jorgensen CM, Hardarson SH, Bek T. The oxygen saturation in retinal vessels from diabetic patients depends on the severity and type of vision-threatening retinopathy. Acta Ophthalmol. 2014 Feb;92(1):34-9. doi: 10.1111/aos.12283. Epub 2013 Dec 16. PMID 24330421
- [Background] Torp TL, Frydkjær-Olsen U, Hansen RS, Peto T, Grauslund J. Intra- and intergrader reliability of semiautomatic measurements of fundus fluorescein angiography leakage in proliferative diabetic retinopathy. European Journal of Ophthalmology, 2015;25(3):e7-e30.
- [Background] Lee CS, Lee AY, Sim DA, Keane PA, Mehta H, Zarranz-Ventura J, Fruttiger M, Egan CA, Tufail A. Reevaluating the definition of intraretinal microvascular abnormalities and neovascularization elsewhere in diabetic retinopathy using optical coherence tomography and fluorescein angiography. Am J Ophthalmol. 2015 Jan;159(1):101-10.e1. doi: 10.1016/j.ajo.2014.09.041. Epub 2014 Oct 25. PMID 25284762
- [Background] de Carlo TE, Bonini Filho MA, Baumal CR, Reichel E, Rogers A, Witkin AJ, Duker JS, Waheed NK. Evaluation of Preretinal Neovascularization in Proliferative Diabetic Retinopathy Using Optical Coherence Tomography Angiography. Ophthalmic Surg Lasers Imaging Retina. 2016 Feb;47(2):115-9. doi: 10.3928/23258160-20160126-03. PMID 26878443
- [Background] Writing Committee for the Diabetic Retinopathy Clinical Research Network; Gross JG, Glassman AR, Jampol LM, Inusah S, Aiello LP, Antoszyk AN, Baker CW, Berger BB, Bressler NM, Browning D, Elman MJ, Ferris FL 3rd, Friedman SM, Marcus DM, Melia M, Stockdale CR, Sun JK, Beck RW. Panretinal Photocoagulation vs Intravitreous Ranibizumab for Proliferative Diabetic Retinopathy: A Randomized Clinical Trial. JAMA. 2015 Nov 24;314(20):2137-2146. doi: 10.1001/jama.2015.15217. PMID 26565927
- [Derived] Vergmann AS, Sorensen KT, Torp TL, Kawasaki R, Wong T, Peto T, Grauslund J. Optical coherence tomography angiography measured area of retinal neovascularization is predictive of treatment response and progression of disease in patients with proliferative diabetic retinopathy. Int J Retina Vitreous. 2020 Nov 4;6(1):49. doi: 10.1186/s40942-020-00249-6. PMID 33292695